CLINICAL TRIAL: NCT06697054
Title: Use of Charcoal Carbon Dye in Sentinel Lymph Node (SLN) Mapping in Early Stage Cervical Cancer
Brief Title: Sentinel Lymph Node (SLN) Mapping with Charcoal Carbon Dye in Early Stage Cervical Cancer
Acronym: SLN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Albayrak, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/1550
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cervical Cancers
Keywords: cervical cancer; indocyanine green; ICG; carbon dye; sentinel lymph node
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: A single arm interventional study aiming at the comparison of the effectiveness of detection for sentinel lymph node biopsy using charcoal carbon dye compared to classic indocyanine (ICG) tracer in early stage cervical cancer.
  Sentinel lymph node detection rates of both tracers in pelvic, obturator and inframesenteric para-aortic whteher bilateral/ unilateral) will be compared in addition to sensitivity, specificity and negative and positive predictive value.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Two different tracers as a sentinel lymph node agent will be compared in early cervical cancer (Experimental): Two different tracers, one charcoal carbon dye and other indocyanine used as sentinel lymph node agent will be compared in early cervical cancer in terms of detection rates, sensitivity, specificity, negative and positive predictive value. Both tracers will be used in the patient.
  Interventions: Diagnostic Test: Sentinel node biopsy with either ICG or carbon dye injection to cervix

INTERVENTIONS:
Diagnostic Test: Sentinel node biopsy with either ICG or carbon dye injection to cervix — Either laparatomy or laparoscopy wil be performed to detect sentinel node stained with either ICG or carbon dye injected to cervix. A hemipelvis in which a sentinel is not found will be subjected to full lymphadenectomy.

SUMMARY:
The aim of the present study is to compare the efficacy of charcoal carbon dye (CCD) in sentinel lymph node mapping compared to indocyanine green (ICG) mapping regarding detection rates, sensitivity, specificity, negative and positive predictive values in early stage cervical cancers (IA2 - IB2).

DETAILED DESCRIPTION:
Cervical cancer continues to be a global health problem despite the advances in prevention, screening and treatment in preinvasive stages. Although radiotherapy is the mainstay of treatment across all stages, surgery with radical and non-radical hysterectomy with pelvic lymph node evaluation is preferred in younger women with early stage cervical cancer who wants to preserve ovarian and sexual functions that may otherwise be hampered by radiotherapy. Lymph node evaluation is critical during and/or after surgery (usually before hysterectomy) and offered by global institutions since hysterectomy during surgery is abandoned in case of a metastasis in pelvic / paraaortic lymph node(s) and/or necessities primary chemoradiation or adjuvant therapy as a therapeutic modality.

During the last 10-15 years surgical sentinel lymph node (SLN) evaluation instead of complete dissection pelvic / paraaortic lymphadenectomy has gained popularity with equal success, especially in cervical tumors with less than 2-4 cm in diameter. Besides, all other advantages of sentinel lymph node evaluation is alike the advantages of other sentinel lymph node evaluation in various other cancers (vulva, breast, endometrial cancers..) with less morbidity such as less vascular injury, lymphedema, lymphocyst formation and etc. Various tracers have been used for sentinel lymph node detection in cervical cancer surgery but indocyanine green (ICG) use has surpassed other SLN mapping tracers and methods and it is the most common agent for detecting SLN in gynecologic oncology. However, it needs a fairly expensive equipment and expertise either by laparoscopy or laparotomy. In the present study, investigators are planning to use charcoal carbon dye (CCD) in addition to ICG as their usual method for SLN mapping. CCD is commonly used by general surgeons for marking of colon during preoperative colonoscopy to delineate the point of resection in surgery for colorectal resection. It is cheap and does not require special equipment and easy to learn. CCD is planned to be given just as the same as giving ICG to the cervix with 1 cc injection at each site of external os (3 and 9 o'clock position, 0.5 cc given to submucosal area and 0.5 given stroma of cervix). 20 minutes following the injection of both agents, laparoscopic dissection of retroperitoneal area will be performed to detect pelvic and paraaortic sentinel lymph nodes (up to inferior mesenteric artery) with ICG and/or CCD.

The aim of the present study is to compare the efficacy of CCD in sentinel lymph node mapping compared to ICG mapping regarding detection rates, sensitivity, specificity, negative and positive predictive values in early stage cervical cancers (IA2 - IB2).

ELIGIBILITY:
Inclusion Criteria: Early stage cervical cancer Stage IA-IB3

-

Exclusion Criteria:

1.Pervious radiotherapy 2.Age less than 18 3.Previous pelvic retroperitoneal surgery

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female (cervical cancer)
Enrollment: 60 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2026-05-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of sentinel lymph node(s) | Two years
  Detection rate of sentinel lymph node(s) either by carbon dye or ICG unilaterally or bilaterally will be recorded and compared.
Specifity of sentinel lymph node mapping by carbon dye or ICG | Two years
  Sensitivities of both tracers for malignancy will be compared to each other
Sensitivity of both tracers will be compared. | Two years
  Sensitivity of both tracers will be compared for malignant metastasis
Sensitivity of both tracers will be compared. | Two years
  Positive and negative predictive values of both tracers for malignant metastasis will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Salihoglu, Prof. Dr., Study Director — ISTANBUL UNİVERSİTY MED FAC DEPT. OF OBSTET AND GYNECOL. DIVISION OF GYNECOLOGİC ONCOLOGY
Locations (1):
- Istanbul University Med Fac Dept. of Obstet and Gynecol. Division of Gynecologic Oncology, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared except personal privacy related ones
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: two years

REFERENCES:
- [Background] ASGE Technology Committee; Kethu SR, Banerjee S, Desilets D, Diehl DL, Farraye FA, Kaul V, Kwon RS, Mamula P, Pedrosa MC, Rodriguez SA, Wong Kee Song LM, Tierney WM. Endoscopic tattooing. Gastrointest Endosc. 2010 Oct;72(4):681-5. doi: 10.1016/j.gie.2010.06.020. PMID 20883844
- [Background] Sun W, Chen X, Fu S, Huang X. Feasibility of Sentinel Lymph Node Mapping With Carbon Nanoparticles in Cervical Cancer: A Retrospective Study. Cancer Control. 2023 Jan-Dec;30:10732748231195716. doi: 10.1177/10732748231195716. PMID 37624147
- [Background] Holloway RW, Abu-Rustum NR, Backes FJ, Boggess JF, Gotlieb WH, Jeffrey Lowery W, Rossi EC, Tanner EJ, Wolsky RJ. Sentinel lymph node mapping and staging in endometrial cancer: A Society of Gynecologic Oncology literature review with consensus recommendations. Gynecol Oncol. 2017 Aug;146(2):405-415. doi: 10.1016/j.ygyno.2017.05.027. Epub 2017 May 28. PMID 28566221
- [Background] Margioula-Siarkou C, Almperis A, Gullo G, Almperi EA, Margioula-Siarkou G, Nixarlidou E, Mponiou K, Papakotoulas P, Sardeli C, Guyon F, Dinas K, Petousis S. Sentinel Lymph Node Staging in Early-Stage Cervical Cancer: A Comprehensive Review. J Clin Med. 2023 Dec 20;13(1):27. doi: 10.3390/jcm13010027. PMID 38202034